CLINICAL TRIAL: NCT04999189
Title: Effectiveness of Using a Mobile Self-care Application in the Management of a Patient With Type 2 Diabetes
Brief Title: The Effectiveness of Using a Mobile Application for Type 2 Diabetes Self-care
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Maribor (Other)
Responsible Party: Principal Investigator, Lucija Gosak, Principal Investigator, University Maribor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 03/5R-2021
Record Dates: First submitted 2021-06-23; First posted 2021-08-10 (Actual); Last update posted 2021-08-10 (Actual); Status verified 2021-08

CONDITIONS: Type 2 Diabetes; Diabetes Mellitus, Type 2; Disease, Chronic; Self-Care; Health Behavior; Mobile Apps; Mobile Phone Use
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Chronic Disease; Health Behavior; Cell Phone Use

STUDY DESIGN:
Masking Description: Masking will not be possible as participants will know to which group they are assigned. The medical staff will also know this as they will teach them how to use the mobile app.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients using mobile applications (Experimental): Patients diagnosed with type 2 diabetes will use a mobile app forDiabetes (Tessera Multimedia, 2020) to manage their disease.
  Interventions: Other: Mobile app forDiabetes (Tessera Multimedia, 2020)
- Control group (No Intervention): Patients will receive treatment from medical staff (as usual).

INTERVENTIONS:
Other: Mobile app forDiabetes (Tessera Multimedia, 2020) — Patients will use a mobile app forDiabetes (Tessera Multimedia, 2020) to manage their disease.
  Arms: Patients using mobile applications

SUMMARY:
The purpose of the research is to evaluate and test the usefulness of the mobile application forDiabetes to improve the self-care of individuals with diabetes type 1. The investigators want to obtain the missing evidence from the field of application operation and their impact on individuals' self-care and study the acceptance of applications among healthcare staff, which plays an essential role in patient education.

DETAILED DESCRIPTION:
The investigators will conduct a randomized study in which individuals included in the intervention group will use the forDiabetes app to self-care for their type 2 diabetes throughout the study. A randomized controlled trial will be conducted in family medicine clinics throughout Slovenia. At the start of the observation and the first control visit, the investigators will assess self-care and disease perception of individuals with the help of validated questionnaires. Measurement of body weight, blood pressure, blood sugar monitoring, and glycated hemoglobin will also be performed at the observation and a first control visit. For individuals who will use the forDiabetes application during the research, the investigators will also assess the frequency of using the mobile application in the home environment at the first control visit.

ELIGIBILITY:
Inclusion Criteria:

* patients older than 18 years;
* with regulated and diagnosed type 2 diabetes;
* patients who are managed in a family medicine clinic;
* patients who have the option of using a mobile phone and a blood sugar meter in the home environment.

Exclusion Criteria:

* patients diagnosed with type 1 diabetes;
* patients who have chronic complications as a result of diabetes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 380 (Estimated)
Dates: Start 2021-09-01 (Estimated); Primary Completion 2022-12-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of change in self-care | up to 6 months
  Self-care in individuals with type 2 diabetes will be assessed using the Self-Care of Diabetes Inventory (SCODI) questionnaire from Ausili et al., 2017. The tool consists of 40 assumptions classified into four dimensions: self-care maintenance (12 assumptions), self-care implementation (8 assumptions), self-care monitoring (9 assumptions), and self-confidence (11 assumptions). The instrument is assessed using the Likert scale, where a higher score represents better self-care.
  Change in SCODI score will be assessed at the enrolment of the patient followed by the examination in the period of up to 6 months after the enrolment.
Assessment of change in disease perception | up to 6 months
  The investigators will use the "Brief Illness Perception Questionnaire" (Brief IPQ) to assess disease perception from authors Broadbent, et al., 2006. The questionnaire provides a rapid assessment of disease perception and measures the patient's cognitive and emotional representations of their disease. The questionnaire contains eight graded questions on a 10-point scale and one open-ended question. The higher the score, the more threatening the individual's view of the disease.
  Change in Brief IPQ score will be assessed at the enrolment of the patient followed by the examination in the period of up to 6 months after the enrolment.
Frequency of using the mobile application | up to 6 months
  The investigators will assess the frequency of use at the first check-up for individuals who will use the application during the research. The questions were partially summarized after the "Video Games Preference Inventory" survey questionnaire from authors Kenny & McDaniel, 2011. In its primary form, the survey questionnaire consists of ten questions. The investigators summarized the first five questions for our research, which the investigators also adapted according to the research content. The questions are rated on the Likert scale (1 = Strongly disagree; 2 = Disagree; 3 = No opinion; 4 = Agree; 5 = Strongly agree). The higher the average rating the user receives, the higher the mobile application level.
  Frequency of the mobile application use will be collected at the examination in the period of up to 6 months after the enrolment.
Change in body weight | up to 6 months
  The registered nurse will measure the patient's body weight with the help of a calibrated technique before the start of the research and at the first examination. The investigators are interested in whether the use of the mobile application will have an effect on weight loss.
Change in glycated hemoglobin | up to 6 months
  The registered nurse will measure the patient's glycated hemoglobin with the help of a calibrated glycated hemoglobin monitor before the start of the research and at the first check-up. The investigators will be able to see if the glycated hemoglobin level has decreased in the time before the examination until the first examination. Recommended target HbA1c is less than 7%.
Change in blood sugar | up to 6 months
  The registered nurse will measure the patient's blood sugar with the help of a calibrated blood sugar monitor before the start of the research and at the first check-up. The investigators will be able to see if the blood sugar level has decreased in the time before the examination until the first examination.
Change in blood pressure | up to 6 months
  The registered nurse will measure the patient's blood pressure with the help of a calibrated blood pressure monitor before the start of the research and at the first check-up. Based on the American Heart Association, these values can be divided into categories (Normal = systolic less than 120, and diastolic less than 80; elevated = systolic between 120 and 129, and diastolic less than 80; hypertension stage 1 = systolic between 130, and 139, or diastolic between 80, and 89; hypertension stage 2 = systolic 140 or higher, or diastolic 90 or higher; hypertension stage 3 = systolic higher than 180, and/or diastolic higher than 120).

CONTACTS AND LOCATIONS:
Overall Officials: Lucija Gosak, Principal Investigator — University of Maribor

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Broadbent E, Petrie KJ, Main J, Weinman J. The brief illness perception questionnaire. J Psychosom Res. 2006 Jun;60(6):631-7. doi: 10.1016/j.jpsychores.2005.10.020. PMID 16731240
- [Derived] Gosak L, Pajnkihar M, Stiglic G. The Impact of Mobile Health Use on the Self-care of Patients With Type 2 Diabetes: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2022 Jun 17;11(6):e31652. doi: 10.2196/31652. PMID 35713944
- See also: Tessera Multimedia, 2020. forDiabetes: diabetes self-management app. [Online] Google Play Store. — https://play.google.com/store/apps/details?id=gr.tessera.fordiabetesapp&hl=en&gl=US
- See also: Ausili, D., et al., 2017. Development and psychometric testing of a theory-based tool to measure self-care in diabetes patients: the Self-Care of Diabetes Inventory. BMC Endocrine Disorders, 17(1), pp. 66. — https://bmcendocrdisord.biomedcentral.com/articles/10.1186/s12902-017-0218-y
- See also: American Heart Association. What do your blood pressure numbers mean? — https://www.heart.org/en/health-topics/high-blood-pressure/understanding-blood-pressure-readings